CLINICAL TRIAL: NCT03460535
Title: Use of the Rhytmia System for Determining the Precise Location and Potential Mechanism of Premature Ventricular Contractions
Brief Title: The Rhytmia System to Determine the Precise Location and Potential Mechanism of Premature Contractions
Acronym: RhytmiaPVC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Boston Scientific Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC31/16/8916; 2017-A00777-46 (Other: ID-RCB)
Record Dates: First submitted 2018-02-26; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Cardiac Arrhythmia; Cardiomyopathy, Dilated
Keywords: Rythmia system
MeSH Terms: conditions — Arrhythmias, Cardiac; Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a purely observational project and the objectives are to record and analyze the local potentials at the site of Premature Ventricular Contraction (VPC) focus through the Rhythmia system, ti determine the short and long-term success of the procedure and compare it to the existing literature about standard procedures, to highlight the advantages of the system compared to conventional mapping and to characterize optimal pace map or activation map as achieved by the Rhythmia system.

DETAILED DESCRIPTION:
This is a purely observational study. No special methodology choice, no comparison.

The study want to find the determination of precise location of the focus and mechanisms involved constitutes a challenge for conventional electrophysiology, even with tridimensional systems, because of the time needed for accurate delineation of the location (due to the sometimes unfrequent Ventricular Premature Beats (VPB)) and to the insufficient mapping density or inadequate signal characteristics. The Rhythmia system could allow better determination of the focus location in relation to the anatomical structures, especially with unfrequent VPB, because of the available high density mapping due to the number of closed high-resolution electrodes located on the Orion catheter. Better delineation of the true focus origin and of the mechanisms involved (automaticity vs re-entry) may be of useful help for better understanding and efficient therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic monomorphic PVC with or without heart disease refractory to anti arrhythmic drugs
* patients with dilated cardiomyopathy and altered Left Ventricular Ejection Fraction (LVEF) suspected to be causes by frequent monomorphic VPC
* patients with malignant ventricular arrhythmias reproducibly induced by monomorphic PVC

Exclusion Criteria:

* patients with non-symptomatic VPC and without cardiomyopathy
* patients under 18 yo
* pregnant women
* patients with polymorphic PVC arising from clearly different areas
* patient protected by the french law: guardianship and Trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited by consultations, hospitalisations or referral by external doctors, in the department of Cardiology.
  This is a purely observational study. No power calculation will be needed due to the lack of comparisons.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Determining the surface of optimal pace map or activation map | One year
  To evaluate the area of isochronal earliest activation of PVC (Premature Ventricular Contraction), based on unipolar or bipolar activation : correlations will be made with the suspected endocardial or epicardial/intra-mural location of the focus. This technic may reduce the area of perfect pace-mapping and possibly more accurately locate the focus.

SECONDARY OUTCOMES:
Record the local potentials at the site of PVC focus through the Rhythmia system | One year
  Pacing from any electrode being in close contact with the endocardial surface and comparing the paced QRS to the spontaneous VPC (automatic calculation available on Bard ElectroPhysiology (EP) system).
  Describe and analyze the local signals recorded from the Orion catheter at the site of the PVC focus.
  by looking for prepotentials as a surrogate of local abnormal automaticity, for local discrete scar and local late potentials favouring local reentry as a cause for PVC, determining the local activation characteristics of VPC (surface of local breakthrough, velocity and direction of activation.
Determine the short success of the procedure | One year
  Determine by repeated Holter recordings, and the relation to the findings made during the procedure (endocardial or suspected epicardial focus), mechanism
Determine long-term success of the procedure and compare it to the existing | One year
  Determine by repeated Holter recordings, and the relation to the findings made during the procedure (endocardial or suspected epicardial focus), mechanism
Characterize optimal pace map or activation map as achieved by the Rhythmia system | One year
  Evaluate the surface of perfect pace-mapping using the Orion catheter, by pacing from any electrode being in close contact with the endocardial surface and comparing the paced QRS to a template of the spontaneous VPC

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Maury, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No